CLINICAL TRIAL: NCT06166901
Title: Evaluation of Long-term Safety and Performance of AcrySof PanOptix Trifocal & PanOptix Toric Trifocal Intraocular Lens (IOLs)
Brief Title: Evaluation of Long-term Safety and Performance of PanOptix Intraocular Lens (IOLs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ILH297-I001
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Aphakia; Astigmatism; Presbyopia
Keywords: Cataract surgery
MeSH Terms: conditions — Aphakia; Astigmatism; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- AcrySof IQ PanOptix IOL - Non Toric (Experimental): Implantation with AcrySof IQ PanOptix non toric IOL in both eyes 3-5 years prior to enrollment
  Interventions: Device: AcrySof IQ PanOptix IOL
- AcrySof IQ PanOptix IOL - Toric (Experimental): Implantation with AcrySof IQ PanOptix IOL in both eyes 3-5 years prior to enrollment, with at least one of the eyes implanted with a toric AcrySof IQ PanOptix IOL
  Interventions: Device: AcrySof IQ PanOptix Toric IOL

INTERVENTIONS:
Device: AcrySof IQ PanOptix IOL — Trifocal IOL implanted in the capsular bag in the eye for the visual correction of aphakia in adult patients with less than 1.00 diopter of preoperative corneal astigmatism, with and without presbyopia, who desire near, intermediate and distance vision with increased spectacle independence.
  Other Names: Model TFNT00
  Arms: AcrySof IQ PanOptix IOL - Non Toric
Device: AcrySof IQ PanOptix Toric IOL — Toric trifocal IOL implanted in the capsular bag in the eye for the visual correction of aphakia and pre-existing corneal astigmatism in adult patients with and without presbyopia, who desire near, intermediate and distance vision with increased spectacle independence.
  Other Names: Models TFNT20, TFNT30, TFNT40, TFNT50, TFNT60
  Arms: AcrySof IQ PanOptix IOL - Toric

SUMMARY:
The purpose of this Post-Market Clinical Follow-up (PMCF) study is to describe the long-term safety and performance of the AcrySof PanOptix Trifocal toric and non-toric IOL models in subjects bilaterally implanted with these IOLs for 3 to 5 years. This study will be conducted in Spain.

DETAILED DESCRIPTION:
Subjects will be recruited from a population that has already undergone lens implantation. Retrospective data will be collected from the pre-operative and surgical visits and any safety outcomes reported prior to enrollment. Prospective data will be collected at Visit 1, which will occur Year 3-5 postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative must be able to understand and sign an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form.
* Subject must have had bilateral implantation of AcrySof PanOptix and/or AcrySof PanOptix Toric IOL models for 3 to 5 years prior to enrollment. A subject may have a Toric lens in one eye and a non-Toric in the fellow eye.
* Subject must have a documented medical history and required pre-operative baseline information available for retrospective data collection.

Exclusion Criteria:

* Subject currently participating in another investigational drug or device study.
* Subject has had corneal refractive surgery after AcrySof PanOptix or AcrySof PanOptix Toric IOL implantation.
* Subject exposed to a study IOL for a minimum of 3 years prior to Visit 1 that have subsequently undergone an IOL exchange and are no longer implanted with a study IOL at the time of enrollment.
* Subject is pregnant or nursing at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Mean Binocular Best Corrected Distance Visual Acuity (BCDVA) | Visit 1 (Year 3-5 postoperative)
  BCDVA will be assessed at a distance of 4 meters using letter charts and recorded in logarithm Minimum Angle of Resolution (logMAR).
Number of Adverse Events (AEs) | Preoperative to Visit 1 (Year 3-5 postoperative)
  Ocular adverse events will be identified from chart review and prospectively at Visit 1. Examples of ocular adverse events include the following:
  * Cystoid Macular Edema (CME)
  * Hypopyon
  * Endophthalmitis
  * Lens dislocation
  * Pupillary block
  * Retinal detachment
  * Secondary Surgical Interventions (explantation/exchange/repositioning)
Number of Device Deficiencies | Preoperative to Visit 1 (Year 3-5 postoperative)
  Device deficiencies will be identified from chart review and prospectively at Visit 1. Examples of device deficiencies include the following:
  * Failure to meet product specifications (e.g., incorrect IOL power)
  * IOL defect
  * Broken IOL optic
  * Broken IOL haptic
  * Scratched IOL optic
  * Unsealed device packaging
  * Suspected product contamination
  * Lack of performance

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research
Locations (7):
- Spain (7):
  - Hospital Universitari General de Catalunya, Sabadell, Barcelona
  - Oftalvist Jerez - HLA Puerta del Sur, Jerez de la Frontera, Cadiz
  - Barraquer Ophthalmology Center, Barcelona
  - Institut Catala de la Retina - Sarria, Barcelona
  - Hospital Arruzafa, Córdoba
  - Miranza IOA, Madrid
  - Clinicas Novovision - Clinica Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No